CLINICAL TRIAL: NCT04612790
Title: A Multinational, Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Investigate the Use of Benralizumab as a Treatment Option for Patients With Bullous Pemphigoid (FJORD)
Brief Title: A Study to Investigate the Use of Benralizumab in Patients With Bullous Pemphigoid.
Acronym: FJORD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Independent Data Monitoring Committee recommended terminating the study following a pre-planned analysis as the efficacy results did not meet the pre-defined futility guidelines. There were no new safety concerns identified from this analysis.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D325AC00002; 2023-505033-27-00 (Other: EU CT); 2020-000287-32 (EudraCT Number)
Record Dates: First submitted 2020-10-12; First posted 2020-11-03 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Bullous Pemphigoid
Keywords: Bullous pemphigoid; rare disease; skin eruptions; itching autoimmune blistering disorder; eosinophilia; urticarial or eczematous or erythematous plaques; bullae; pruritus
MeSH Terms: conditions — Pemphigoid, Bullous; Rare Diseases; Eosinophilia; Urticaria; Blister; Pruritus | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab (Experimental): Benralizumab subcutaneously (SC) loading dose followed by repeat dosing of SC benralizumab plus Oral Corticosteroids per SoC tapering.
  Open-Label (OLE): after completion of the double-blind treatment period, all participants will have the option of entering an OLE period, starting at week 36 benralizumab SC until study closure.
  Interventions: Biological: Benralizumab
- Placebo (Experimental): Placebo plus Oral Corticosteroids per SoC tapering. Open-Label (OLE): after completion of the double-blind treatment period, all participants will have the option of entering an OLE period, starting at week 36 benralizumab SC until study closure.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab subcutaneously (SC) loading dose followed by repeat dosing of SC benralizumab plus Oral Corticosteroids per SoC tapering.
  Open-Label (OLE): after completion of the double-blind treatment period, all participants will have the option of entering an OLE period, starting at week 36 benralizumab SC until study closure.
  Other Names: Benralizumab, Benra, Fasenra
  Arms: Benralizumab
Biological: Placebo — Placebo plus Oral Corticosteroids per SoC tapering. Open-Label (OLE): after completion of the double-blind treatment period, all participants will have the option of entering an OLE period, starting at week 36 benralizumab SC until study closure.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the use of benralizumab is effective in the treatment of patients symptomatic Bullous Pemphigoid (BP).

DETAILED DESCRIPTION:
Bullous pemphigoid (BP) is a rare disease mainly affecting the elderly. BP is associated with significant morbidity and increased mortality secondary to increased risk of secondary infections, comorbid conditions, and serious side effects from high-dose steroids and immunosuppressants. The aim of this study is to investigate the use of benralizumab as a treatment for patients symptomatic with Bullous Pemphigoid (BP).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Informed Consent/Age

1. Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
2. Adult participants ≥ 18 years of age at the time of signing the ICF.

   Type of Participant and Disease Characteristics
3. Participants must have clinical features of BP (eg, urticarial or eczematous or erythematous plaques, bullae, pruritus) at the screening visit and confirmed diagnosis with histology, direct immunofluorescence, and serology at randomization. Required for inclusion:

   1. Histology.
   2. Positive direct immunofluorescence (from skin biopsy) (IgG and/or C3 at the basement membrane zone).
   3. AND at least one of the following serologic assessments positive (all assessed from participant's blood sample):

   (i) indirect immunofluorescence (IgG on the roof of salt- split skin). (ii) positive serology on ELISA for BPAG1 (230-kd). (iii) positive serology on ELISA for BPAG2 (180-kd).
4. BPDAI activity score ≥ 24 at the screening and randomization visits.
5. Candidate for systemic corticosteroid therapy.
6. Able to complete PRO assessments on a tablet and on a handheld device. Some participants may be exempted from completing home PROs on the handheld device upon agreement with the AstraZeneca physician (eg, if the patient has a medical condition such as BP lesions of the fingers/hand, a neurologic condition affecting fingers/hand, or severe visual impairment).

Sex 7 Male or female.

Reproduction 8 Female participants capable of having children must meet both of the following conditions ([a] and [b]):

(a) Have a negative urine pregnancy test at screening and (b) Must agree to use a highly effective method of birth control (confirmed by the investigator) from randomization throughout the study duration and within 12 weeks after last dose of IP. Highly effective forms (those that can achieve a failure rate of less than 1% per year when used consistently and correctly) of birth control include: (i) Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation - oral, intravaginal, or transdermal.

(ii) Progestogen-only hormonal contraception associated with inhibition of ovulation - oral, injectable, or implantable.

(iii) Intrauterine device. (iv) Intrauterine hormone-releasing system. (v) Bilateral tubal occlusion. (vi) Sexual abstinence, ie, refraining from heterosexual intercourse (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant).

(vii) Vasectomized sexual partner provided that partner is the sole sexual partner of the female of childbearing potential (FOCBP) study participant and that the vasectomized partner has received medical assessment of the surgical success.

(c) Females not of childbearing potential are defined as females who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Females will be considered postmenopausal if they have been amenorrhoeic for ≥ 12 months prior to the planned date of randomization without an alternative medical cause. The following age-specific requirements apply: (i) Females < 50 years old will be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and follicle-stimulating hormone (FSH) levels in the postmenopausal range. Until FSH is documented to be within menopausal range, treat the participant as a female of childbearing potential.

(ii) Females ≥ 50 years old will be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatment.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Forms of BP other than classic, predominantly cutaneous BP: eg, mucous membrane BP, epidermolysis bullosa acquisita, Brunsting-Perry BP, p200 BP, p105 BP, BP with concomitant pemphigus vulgaris, and drug-induced BP.
2. Comorbid disease that in the Investigator's judgement might interfere with the evaluation of the IP or safety of the participant. This includes any disorder that in the opinion of the Investigator is not stable (eg, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment).
3. Current or history of malignancy within 5 years before the screening visit with the following exceptions:

   1. Participants treated for in situ carcinoma of the cervix who have completed curative therapy and are in remission for at least 12 months prior to signing the informed consent and
   2. Participants with superficial basal cell or squamous skin cancer.
   3. Participants who have had other malignancies are eligible provided that the participant is in remission and curative therapy was completed at least 5 years prior to the date informed consent was obtained.
4. History of anaphylaxis to any biologic therapy or vaccine.
5. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy.
6. Any clinically significant abnormal findings in physical examination, vital signs, electrocardiogram (ECG), hematology, or clinical chemistry during screening, which in the opinion of the Investigator, may put the participant at risk because of his/her participation in the study, or may influence the results of the study.
7. Current active liver disease.

   1. Chronic stable hepatitis B and C (including positive testing for hepatitis B surface antigen or hepatitis C antibody), or other stable chronic liver disease are acceptable if participant otherwise meets eligibility criteria. Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice, or cirrhosis.
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥3 times the upper limit of normal, confirmed by repeated testing during screening period. Transient increase of AST/ALT level that resolves by the time of randomization is acceptable if in the Investigator's opinion the participant does not have an active liver disease and meets other eligibility criteria.
8. A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test.

   Prior/Concomitant Therapy
9. Use of immunosuppressive medication, including, but not limited to: methotrexate, cyclosporine, azathioprine, within 4 weeks or 5 half-lives prior to the date informed consent is obtained, whichever is longer.

   Other Exclusions
10. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained.
11. Receipt of any marketed or investigational biologic within 4 months or 5 half-lives prior to the date informed consent is obtained, whichever is longer. Participants on stable therapy for at least 3 months before randomization who intend to stay on treatment throughout the study with marketed biologics that are not likely to interfere with the assessment of safety and/or efficacy of benralizumab (eg, for the treatment of osteoporosis, migraine, pain, diabetes, obesity, ocular, cardiovascular, or metabolic diseases) can participate in the study.
12. Known history of allergy or reaction to any component of the IP formulation.
13. Receipt of live attenuated vaccines 30 days prior to the date of randomization.
14. Previously received benralizumab (MEDI-563, FASENRA).
15. Change to allergen immunotherapy or new allergen immunotherapy within 30 days prior to the date of informed consent and anticipated changes in immunotherapy throughout the study.
16. Planned elective major surgical procedures during the conduct of the study.
17. Previous randomization in the present study.
18. Concurrent enrollment in another interventional (eg, investigational drug or device) clinical trial.
19. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
20. For females only: Currently pregnant, breastfeeding, or lactating females.

    (a) A urine pregnancy test must be performed for FOCBP at Visit 1. A positive urine test result must be confirmed with a serum pregnancy test. If serum test is positive, the participant should be excluded.
21. Participant is unable to complete PRO assessments because of cognitive function (eg, dementia).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (6):
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Centennial, Colorado
  - Research Site, Margate, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Beverly, Massachusetts
- Australia (3):
  - Research Site, Kogarah
  - Research Site, Parkville
  - Research Site, Westmead
- Bulgaria (2):
  - Research Site, Haskovo
  - Research Site, Sofia
- China (4):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Hohhot
  - Research Site, Shanghai
- France (4):
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Rouen
- Germany (4):
  - Research Site, Bad Bentheim
  - Research Site, Bielefeld
  - Research Site, Dresden
  - Research Site, Leipzig
- Research Site, Thessaloniki, Greece
- Israel (2):
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (3):
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Rome
- Japan (7):
  - Research Site, Iruma-Gun
  - Research Site, Kitakyusyu-shi
  - Research Site, Kurume-shi
  - Research Site, Okayama
  - Research Site, Ōta-ku
  - Research Site, Sapporo
  - Research Site, Urayasu-shi
- Spain (2):
  - Research Site, Alicante
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: FJORD Brochure — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D325AC00002&attachmentIdentifier=3b7a1bd4-a4a0-42a3-8005-b752575578aa&fileName=Fjord_Brochure_DL_8pg_V02.pdf&versionIdentifier=
- See also: FJORD Flyer — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D325AC00002&attachmentIdentifier=7b27b1f1-8cac-44ff-8ead-d4df5313b50f&fileName=FJORD_Flyer_V01_Global(en).pdf&versionIdentifier=
- See also: A website on the FJORD study. — https://www.astrazenecaclinicaltrials.com/study/D325AC00002/
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D325AC00002&attachmentIdentifier=83c52916-ce4a-41c7-bd35-826114393df6&fileName=d325ac00002-synopsis_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in adult participants with symptomatic bullous pemphigoid (BP) at 32 sites in 11 countries. Study consisted of screening period, double-blind (DB) period in which 67 participants were randomized in 1:1 ratio to either receive benralizumab or placebo for 36 weeks followed by optional open-label extension (OLE) period (for participants who completed the DB period), in which all participants received benralizumab for at least 1 year.
Pre-assignment Details: Study was terminated following a pre-planned futility analysis as efficacy results did not pass pre-defined futility hurdle. Prior to futility analysis,AstraZeneca created protocol#5 and Statistical analysis plan(SAP)#3. Updated protocol was never submitted to health authorities as study was terminating. Results align with protocol#5 and SAP#3.
Groups:
- DB Period: Benralizumab: Participants received benralizumab with an initial loading dose of 60 milligrams (mg) followed by a maintenance dose of 30 mg every 4 weeks (Q4W) as a subcutaneous (SC) injection for 36 weeks.
- DB Period: Placebo: Participants received volume-matched placebo as a SC injection on the same dosing schedule as benralizumab Q4W for 36 weeks.
- OLE Period: Benralizumab (DB)/Benralizumab (OLE): Participants who received benralizumab in DB period received benralizumab 30 mg Q4W in OLE period for at least 1 year.
- OLE Period: Placebo (DB)/Benralizumab (OLE)-: Participants who received matched placebo in DB period received benralizumab 30 mg Q4W in OLE period for at least 1 year.
Period: DB Period (Up to 36 Weeks)
Arm/Group | DB Period: Benralizumab | DB Period: Placebo | OLE Period: Benralizumab (DB)/Benralizumab (OLE) | OLE Period: Placebo (DB)/Benralizumab (OLE)-
Started | 34 | 33 | 0 | 0
Completed | 16 | 19 | 0 | 0
Not Completed | 18 | 14 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 8 | 6 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 0 | 0
Not completed — Physician Decision | 4 | 3 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0
Period: OLE Period (Up to 1 Year)
Arm/Group | DB Period: Benralizumab | DB Period: Placebo | OLE Period: Benralizumab (DB)/Benralizumab (OLE) | OLE Period: Placebo (DB)/Benralizumab (OLE)-
Started | 0 | 0 | 16 | 18
Randomized But Did Not Receive Treatment in OLE Period | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 16 | 18
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Investigator decision | 0 | 0 | 2 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 14 | 15
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of investigational product (IP), irrespective of their protocol adherence and continued participation in the study.
Groups:
- DB Period: Benralizumab: Participants received benralizumab with an initial loading dose of 60 mg followed by a maintenance dose of 30 mg Q4W as a SC injection for 36 weeks.
- Total: Total of all reporting groups
Arm/Group | DB Period: Benralizumab | DB Period: Placebo | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (10.4) | 72.5 (11.4) | 70.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 14 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 34 | 32 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 13 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 16 | 20 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders at Week 36
Description: A responder was defined as a participant who was in complete remission while off OCS for ≥2 months at Week 36.
Time Frame: At Week 36
Population: FAS included all randomized participants who received at least 1 dose of IP, irrespective of their protocol adherence and continued participation in the study. Only participants who had the opportunity to reach Week 36 are included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DB Period: Benralizumab | DB Period: Placebo
Number analyzed (Participants) | 18 | 19
Percentage of participants | 11.1 [-2.70 to 26.11] | 5.26 [-5.06 to 15.07]
Statistical Analysis 1: Comparison: DB Period: Benralizumab vs DB Period: Placebo; Estimates were from a logistic regression model using the Firth adjustment (adj) that included treatment group, baseline disease severity (moderate, severe) and time of BP diagnosis (participants with newly diagnosed BP, participants with a previous diagnosis of BP who have relapsed) as categorical covariates; Test type: Other; p = 0.509, Logistic regression model with Firth adj; Difference in percentage of responders = 6.70, 95% CI 2-sided [-10.90 to 24.29]

2. Secondary Outcome: Percentage of Participants Who Remained Relapse-Free up to Week 36
Description: Relapse was defined as the appearance of 3 or more new lesions per month (blisters, eczematous lesions, or urticarial plaques); or at least 1 large (>10 centimeter [cm] diameter) eczematous lesion or urticarial plaques that did not heal within 1 week; or the extension of established lesions or daily pruritus in participants who had achieved disease control.
Time Frame: Up to Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DB Period: Benralizumab | DB Period: Placebo
Number analyzed (Participants) | 18 | 19
Percentage of participants | 23.78 [5.95 to 41.61] | 19.79 [1.43 to 38.15]

3. Secondary Outcome: Cumulative OCS Exposure From Baseline to Week 36
Description: The cumulative OCS exposure was estimated as the sum over the relevant 4-week periods from the mixed-effect model for repeated measures (MMRM) model. Baseline was defined as the last recorded value on or prior to the date of randomization. Equivalents were prednisone equivalents (converted from mg).
Time Frame: Baseline (Day 1) and Week 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg per kilogram (mg/kg)
Arm/Group | DB Period: Benralizumab | DB Period: Placebo
Number analyzed (Participants) | 18 | 19
mg per kilogram (mg/kg) | 71.37 (63.19) | 62.71 (46.90)

4. Secondary Outcome: Change From Baseline in Bullous Pemphigoid Disease Area Index (BPDAI) Activity Score at Week 36
Description: BPDAI is a clinician completed tool that is used for independent disease severity assessment to measure disease extent in BP. The total BPDAI activity score is calculated as the arithmetic sum of the 3 subcomponents - cutaneous blisters/erosions, cutaneous urticaria/erythema, and mucosal blisters/erosions. The BPDAI total activity gives an indication of disease activity, with score range from 0 (no disease activity) to 360 (severe disease activity). Higher scores indicating greater disease activity. Baseline was defined as the last recorded value on or prior to the date of randomization.
Time Frame: Baseline (Day 1) and Week 36
Population: FAS included all randomized participants who received at least 1 dose of IP, irrespective of their protocol adherence and continued participation in the study. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DB Period: Benralizumab | DB Period: Placebo
Number analyzed (Participants) | 14 | 12
Score on a scale | -53.29 (46.33) | -52.75 (17.36)

5. Secondary Outcome: Change From Baseline in BPDAI-Pruritus Score at Week 36
Description: The BPDAI-Pruritus is a separate component of the BPDAI that asks the participant to grade the severity of pruritus over the past 24 hours, the past week, and the past month. For each recall period, severity of pruritus is rated on a numeric rating scale (NRS) ranging from 0 for no itch to 10 for maximal itching. The BPDAI-Pruritus score was computed as the sum of 3 components ranging from 0 to 30. Higher scores indicated worse condition. Baseline was defined as the last recorded value on or prior to the date of randomization.
Time Frame: Baseline (Day 1) and Week 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DB Period: Benralizumab | DB Period: Placebo
Number analyzed (Participants) | 14 | 12
Score on a scale | -5.57 (7.23) | -16.58 (9.21)

6. Secondary Outcome: Cumulative OCS Exposure From Baseline to Week 16
Description: The cumulative OCS exposure was estimated as the sum over the relevant 4-week periods from the MMRM model. Baseline was defined as the last recorded value on or prior to the date of randomization. Equivalents were prednisone equivalents (converted from mg).
Time Frame: Baseline (Day 1) and Week 16
Population: FAS included all randomized participants who received at least 1 dose of IP, irrespective of their protocol adherence and continued participation in the study. Only participants who had the opportunity to reach Week 16 are included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | DB Period: Benralizumab | DB Period: Placebo
Number analyzed (Participants) | 24 | 24
mg/kg | 46.90 (27.19) | 42.15 (33.33)

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious AEs were collected from first dose of study treatment (Day 1) up to study termination (approximately 133 weeks).
Description: The safety analysis set consists of all participants who had received at least 1 dose of IP.
Groups:
- OLE Period: Placebo (DB)/Benralizumab (OLE): Participants who received matched placebo in DB period benralizumab 30 mg Q4W in OLE period for at least 1 year.
Arm/Group | DB Period: Benralizumab | DB Period: Placebo | OLE Period: Benralizumab (DB)/Benralizumab (OLE) | OLE Period: Placebo (DB)/Benralizumab (OLE)
All-Cause Mortality (participants affected / at risk) | 1/34 | 1/33 | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 9/34 | 8/33 | 4/16 | 2/18
Other Adverse Events (participants affected / at risk) | 22/34 | 23/33 | 8/16 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Benralizumab (N=34) | DB Period: Placebo (N=33) | OLE Period: Benralizumab (DB)/Benralizumab (OLE) (N=16) | OLE Period: Placebo (DB)/Benralizumab (OLE) (N=18)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Benralizumab (N=34) | DB Period: Placebo (N=33) | OLE Period: Benralizumab (DB)/Benralizumab (OLE) (N=16) | OLE Period: Placebo (DB)/Benralizumab (OLE) (N=18)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 6 (6) | 4 (4) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 1 (2)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (4) | 1 (1)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (5) | 2 (2) | 1 (1) | 1 (1)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated following a pre-planned futility analysis as the efficacy results did not pass the pre-defined futility hurdle with no new safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT04612790/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT04612790/SAP_001.pdf